CLINICAL TRIAL: NCT03731858
Title: Role of HbA1c in Intracytoplasmic Sperm Injection
Brief Title: HbA1c in Intracytoplasmic Sperm Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ICSI
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ICSI has increased nowadays for treating cases of longstanding infertility . HbA1c has an important value in evaluating glucose level in blood

DETAILED DESCRIPTION:
- The level of HbA1c in blood denotesnthe glycemic control over the past 3 months . Its regulation is very important in human reproductive life

ELIGIBILITY:
Inclusion Criteria:

* females with infertility from 20 to 42 years old

Exclusion Criteria:

* females with age below 20 or above 42 years

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile ladies
Study Population: -Any lady with infertilty and has a recurrent ICSI trials
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
the number of ladies who will get pregnant | within one year
  the ladies who will become pregnant after ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt